CLINICAL TRIAL: NCT05812469
Title: The Effect of a Psychoeducational Intervention for Brain Awareness Applied on Patients With Alcohol and Substance Use Disorders on Metacognition, Self-efficacy and Treatment Motivation
Brief Title: A Psychoeducational Intervention for Brain Awareness, Metacognition, Self-efficacy and Treatment Motivation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Halil İbrahim ÖLÇÜM, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BA-project
Record Dates: First submitted 2023-03-01; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Substance Use Disorders; Alcohol Use Disorder
Keywords: Brain Awareness; Psychoeducation; Metacognition; Self-efficacy; Treatment Motivation
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism

STUDY DESIGN:
Intervention Model Description: It is an experimentally designed study with a randomized control group and repeated measurements (pre-test, mid-test, post-test).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): psychoeducation and counseling provided as part of the Brain Awareness Intervention for the experimental group of 39 patients
  Interventions: Behavioral: Brain Awareness Intervention
- control group (Active Comparator): 38 patients will receive education about Being Healthy
  Interventions: Behavioral: Being Healthy Education

INTERVENTIONS:
Behavioral: Brain Awareness Intervention — effect of brain awareness intervention on metacognition, self-efficacy and treatment motivation in patients with alcohol and substance use disorders
  Arms: experimental group
Behavioral: Being Healthy Education — This training included trainings on Healthy Nutrition, Sexually Transmitted Diseases, Importance of Physical Activity and Personal Hygiene prepared by the researcher in the form of presentations for the patients in the control group.
  Arms: control group

SUMMARY:
The aim of this study is to examine the effect of brain awareness intervention on metacognition, self-efficacy and treatment motivation in patients with alcohol and substance use disorders. It is an experimentally designed study with a randomized control group and repeated measurements (pre-test, mid-test, post-test).

DETAILED DESCRIPTION:
The aim of this study is to examine the effect of brain awareness intervention on metacognition, self-efficacy and treatment motivation in patients with alcohol and substance use disorders. It is an experimentally designed study with a randomized control group and repeated measurements (pre-test, mid-test, post-test). 77 inpatients at the Alcohol and Drug Addiction Treatment and Research Center included between April and October 2021. In addition to standard treatment, psychoeducation and counseling provided as part of the Brain Awareness Intervention for the experimental group of 39 patients. The control group of 38 patients will receive education about Being Healthy in addition to standard treatment and standard follow-up. Patients' pathological metacognitive activities, self-efficacy perceptions and treatment motivation will assessed with the Metacognition Scale-30, Self-Efficacy Scale and Treatment Motivation Questionnaire using one-way and two-way repeated measures analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Being between the ages of 18-65 and able to read and write
2. Inpatient treatment with alcohol or substance abuse problem
3. To not have a psychiatric (severe depression, bipolar disorder or psychosis) or mental illness that would prevent participation in the study

Exclusion Criteria:

1. Failure to participate in more than one session despite agreeing to participate in the research
2. Taking the decision to terminate treatment or early discharge by violating treatment rules during the treatment process
3. Not participating in post-discharge follow-up or post-test application

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Metacognition Scale-30 | 72 Hours
  There are five sub-factors of the PPI-30 scale: Positive beliefs (items 1,7,10,20,23 and 28), Uncontrollability and danger (items 2,3,4,9,11,16 and 22), Cognitive confidence (items 8,14,18,24,26 and 29), Need to control thoughts (items 6,13,15,21,25 and 27) and Cognitive awareness (items 5,12,17,19 and 30).
  The PPI-30 is a four-point Likert-type scale ranging from "1 - Strongly disagree" to "4 - Strongly agree". Scores between 30 and 120 can be obtained from the scale, there is no reverse-scored item, and a higher score indicates an increase in pathological metacognitive activity. It is reported that the Cronbach Alpha reliability value of the Turkish version of the scale is 0.86 and the Cronbach Alpha value of the sub-dimensions is between 0.72 and 0.93.
Self-Efficacy-Efficacy Scale | 72 Hours
  The 23-question form of the scale has four subscales: initiating the behavior, maintaining the behavior, completing the behavior and struggling with obstacles.
  The SCBS is a five-point Likert-type scale ranging from "1 - does not describe me at all" to "5 - describes me very well". Scores between 23 and 115 can be obtained from the scale. Items 2,4,5,6,7,10,11,12,12,14,16,17,18,20 and 22 in the scale are reverse-scored and an increase in the total score means that the individual's self-efficacy perception is at a good level. The Cronbach Alpha reliability value of the Turkish version of the scale is 0.81.
Treatment Motivation Questionnaire | 72 Hours
  The Treatment Motivation Questionnaire is a five-point Likert-type questionnaire ranging from "1 - Strongly disagree" to "5 - Strongly agree". A score between 26-130 can be obtained from the questionnaire. Items 13, 16, 21 and 24 in the questionnaire are reverse-scored in the opposite direction and an increase in the total score obtained from the questionnaire means that the individual's treatment motivation is high. The Cronbach Alpha reliability value of the Turkish version of the questionnaire is 0.84.

CONTACTS AND LOCATIONS:
Locations (1):
- Halil Ibrahim Olcum, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No